CLINICAL TRIAL: NCT02586311
Title: A Randomized, Double-blind, Multi-center, Phase 3 Trial to Evaluate the Efficacy and Safety of a CKD-330 Versus Amlodipine Monotherapy in Hypertensive Patients Inadequately Controlled by Amlodipine Monotherapy
Brief Title: CKD-330 Phase 3 Trial in Amlodipine Non-responder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 144HT15027
Record Dates: First submitted 2015-10-23; First posted 2015-10-26 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Amlodipine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CKD-330 16/5mg + Amlodipine 5mg placebo (Experimental): CKD-330 16/5mg + Amlodipine 5mg placebo, po, q.d.
  Interventions: Drug: CKD-330 16/5mg; Drug: Amlodipine 5mg Placebo
- CKD-330 16/5mg placebo + Amlodipine 5mg (Active Comparator): CKD-330 16/5mg placebo + Amlodipine 5mg, po, q.d.
  Interventions: Drug: CKD-330 16/5mg Placebo; Drug: Amlodipine 5mg

INTERVENTIONS:
Drug: CKD-330 16/5mg — Once a day, 8 weeks
  Arms: CKD-330 16/5mg + Amlodipine 5mg placebo
Drug: Amlodipine 5mg Placebo — Once a day, 8 weeks
  Other Names: Norvasc 5mg Placebo
  Arms: CKD-330 16/5mg + Amlodipine 5mg placebo
Drug: CKD-330 16/5mg Placebo — Once a day, 8 weeks
  Arms: CKD-330 16/5mg placebo + Amlodipine 5mg
Drug: Amlodipine 5mg — Once a day, 8 weeks
  Other Names: Norvasc 5mg
  Arms: CKD-330 16/5mg placebo + Amlodipine 5mg

SUMMARY:
Trial to Evaluate the Efficacy and Safety of a CKD-330 versus Amlodipine Monotherapy in Hypertensive Patients Inadequately Controlled by Amlodipine Monotherapy

DETAILED DESCRIPTION:
A Randomized, Double-blind, Multi-center, Phase 3 Trial to Evaluate the Efficacy and Safety of a CKD-330 versus Amlodipine Monotherapy in Hypertensive Patients Inadequately Controlled by Amlodipine Monotherapy

ELIGIBILITY:
Inclusion Criteria:

* Age of 19 or above
* Essential hypertension with 140mmHg ≤ mean sitSBP < 180mmHg on target arm at Visit 2
* Ability to provide written informed consent

Exclusion Criteria:

* The difference between arms of sitSBP ≥ 20mmHg and/or sitDBP ≥ 10mmHg at Visit 1
* mean sitSBP ≥ 200mmHg and/or mean sitDBP ≥ 120mmHg on target arm at Visit 1
* mean sitSBP ≥ 180mmHg and/or mean sitDBP ≥ 120mmHg on target arm at Visit 2
* Known or suspected Secondary Hypertension
* Type I Diabetes Mellitus and Type II Diabetes Mellitus with HbA1c > 9%
* Patients with severe congestive heart failure(NYHA class III, IV)
* Patient with ischemic heart disease, Ischemic cardiovascular disease, Valvular heart disease, arrhythmia requiring treatment within 3 months
* History of cerebrovascular disease as cerebral infarction, cerebral hemorrhage within 6 months
* History of severe or malignant retinopathy
* AST/ALT ≥ UNL*3, Serum creatinine ≥ UNL*1.5, K > 5.5mEq/L
* Patients with acute or chronic inflammatory status requiring treatment
* Patient who need to take antihypertensive drug besides Investigational products
* Patient must be treated with medications prohibited for concomitant use during the study period
* History of angioedema related to ACE inhibitor or angiotensin II receptor blockers
* History of disability to drug ADME, active inflammatory bowel syndrome within 12months, impaired pancreatic function, GI bleeding, obstructions of urinary tract
* History of malignant tumor within 5 years
* Patient who are dependent on drugs or alcohol within 6 months
* Hypersensitive to Candesartan/Amlodipine
* Women with pregnant, breast-feeding
* Patients treated with other investigational product within 30 days at first time taking the investigational product
* Not eligible to participate for the study at the discretion of investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2016-01; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
The mean change of sitSBP(sitting Systolic blood pressure) | From baseline at week 8

SECONDARY OUTCOMES:
The mean change of sitSBP(sitting Systolic blood pressure) | From baseline at week 4
The mean change of sitDBP(sitting diastolic blood pressure) | From baseline at week 4 and week 8
Blood Pressure Control rate | From baseline to week 8
  Patient achieving sitSBP < 140mmHg and sitDBP < 90mmHg
Blood Pressure Response rate | From baseline to week 8
  sitSBP reduction ≥ 20mmHg and sitDBP reduction ≥ 10mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Chang Gyu Park, M.D, Ph.D, Principal Investigator — Korea University Guro Hospital
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No